CLINICAL TRIAL: NCT04954235
Title: Effectiveness and Safety Study of Specific Hyperimmune Equine Serum for the Treatment of Severe Hospitalized SARS-CoV-2 in Adults: Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Inmunova S.A. (Other)
Collaborators: Hospital Italiano de Buenos Aires (Other); Hospital de Campaña Escuela Hogar (Unknown); Laboratorio Elea Phoenix S.A. (Industry); Instituto de Virologia Dr. Jose Maria Vanella (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4484
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to Anti-SARS-CoV-2 hyperimmune equine immunoglobulin F[ab']2 fragments: Group of patients with severe pneumonia who received treatment with 2 infusions of 4 mg / Kg each of hyperimmune anti-SARS-CoV-2 serum (INM005, CoviFab®) separated by 48 hours
- Not Exposed to Anti-SARS-CoV-2 hyperimmune equine immunoglobulin F[ab']2 fragments: Group of patients with severe pneumonia not exposed to hyperimmune anti-SARS-CoV-2 serum (INM005, CoviFab®) during hospitalization corresponding to the period prior to the approval of the hyperimmune anti-SARS-CoV-2 serum for its use.

SUMMARY:
An observational, retrospective, classic cohort study of adult patients hospitalized for severe pneumonia with a diagnosis of SARS-CoV-2 by RT-PCR will be carried out. The cohort will be divided into two arms: a group of patients who received treatment with anti-SARS-CoV-2 hyperimmune serum and a group of patients not exposed to the intervention during hospitalization corresponding to the period prior to the approval of the anti-hyperimmune serum SARS-CoV-2 for use. All patients will be have structured follow-up at 14, 21 and 28 days, until discharge or death.

DETAILED DESCRIPTION:
A classic retrospective cohort observational study of adult patients hospitalized for severe pneumonia with a diagnosis of SARS-CoV-2 will be conducted. The date of admission to the cohort will be considered the date of admission. All patients will be followed with structured evaluations at 14, 21 and 28 days.

The cohort will be divided into two arms: a group of patients who received treatment with 2 infusions of 4 mg / Kg each of hyperimmune anti-SARS-CoV-2 serum (INM005, CoviFab®) separated by 48 hours, from the date of approval for its use; and a group of patients not exposed to said intervention during hospitalization corresponding to the period prior to the approval of the hyperimmune anti-SARS-CoV-2 serum for its use. CoviFab® has been authorized under special conditions by the Agency for Medicines, Food and Medical Technology (ANMAT) for the treatment of hospitalized patients with moderate to severe disease caused by the SARS-CoV-2 virus (Regulation 9175/20, 22 December 2020)

The study period that will be considered for the arm of patients exposed to anti-SARS-CoV-2 polyclonal hyperimmune serum is between January 27, 2021 and April 9, 2021. The study period to include patients not exposed to hyperimmune anti-SARS-CoV-2 serum is between September 1, 2020 to January 26, 2021. This last period was chosen because it is considered to be a time when there were no substantive differences in the diagnosis, categorization of risk, support measures or treatment of hospitalized adult patients with a confirmed diagnosis of COVID-19 pneumonia, and therefore corresponds to a valid period for comparison.

Although the "Escuela Hogar" Hospital began operating in July 2020, it was decided to exclude patients admitted for the first two months, considering that after two months of operation, the diagnostic, treatment and support systems are stable for the comparison between exposed and unexposed patients.

The study will be carried out in a collaborative manner between the Acute Campaign Hospital "Escuela Hogar" and the Hospital Italiano de Buenos Aires, which will act as the coordinating center for this study.

The Acute Campaign Hospital "Escuela Hogar" was designed and implemented to treat COVID-19 cases exclusively. It was inaugurated in July 2020 in the city of Corrientes, Argentine Republic, with the aim of functioning as a diagnostic and treatment center for patients affected by COVID-19 throughout the province of Corrientes[4].

It has a general hospitalization sector and a intensive care unit, with approximately 723 total beds available and 300 in the intensive care unit. The staff includes doctors, nurses and health personnel, as well as technicians and administrators trained in the care of patients affected by COVID-19. It has an Operations Center where the members of the Crisis Committee monitor the entire building and access in real time, the status of patients and the movement of that institution.

The hospital is paper free, and has a Computerized Medical Record. This data repository has additional information on patient admission, free text evolutions, structured indications, vital sign registration and support, and results of imaging studies reports such as X-rays and Tomography. The laboratory is in a different development that contains all the laboratories performed on each patient in each episode.

The data processing and analysis will be carried out in the area of the Research Department of the Hospital Italiano de Buenos Aires.

Variables Follow-up will be carried out with structured forms upon admission, days 14, 21 and 28. For the purposes of the study, we will include demographic variables (age, sex, BMI), presence of comorbidities (hypertension, diabetes, obesity, cancer, lung disease, liver disease, kidney disease, coronary / cardiovascular disease), the history of having received plasma in the previous 30 days or during hospitalization, the plasma dose, Charlson score; related to the patient's diagnosis and their baseline status at admission (diagnostic method , date of onset of symptoms, respiratory rate, oxygen saturation, PaO2 / FiO2, oxygen requirement, type of device indicated, NEWS score) and related to the evolution both in hospitalization and after hospital discharge until day 28 from hospital admission (need for supplemental oxygen, admission to mechanical ventilation, admission to ICU, clinical improvement, disease progression, death, discharge).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and younger than 80 years.
* Hospitalized for COVID-19 at the "Escuela Hogar" Hospital in Corrientes, Argentina from September 2020 to April 2021.
* Confirmed diagnosis of COVID-19 by SARS-CoV-2 Antigen Test or qualitative reverse transcriptase-polymerase chain reaction (qRT-PCR -GeneoDX Co, Ltd or similar) or Dosage of anti-SARS-CoV-2 IgG / IgM antibodies
* Who received hyperimmune anti-SARS-CoV-2 serum according to the indication approved by ANMAT for use after the approval date (January 2021 to April 2021) or Patients with the same indication corresponding to the period prior to the approval date (September 2020 to January 2020)
* With severe disease defined as individuals with tachypnea> 30 breaths per minute or oxygen saturation <94% ambient air or PaO2 / FiO2 <300, or pulmonary infiltrates> 50% on chest image.

Exclusion Criteria:

* Asymptomatic disease (individuals with a positive test for SARS-CoV-2, but who do not have symptoms), mild (individuals who have compatible symptoms, but without dyspnea and with a normal chest imaging study), moderate (individuals with evidence of lower respiratory tract disease on clinical or imaging evaluation, and oxygen saturation> = 94% room air) or critical (those with respiratory failure, septic shock, and / or multi-organ dysfunction).
* Patients who received anti-SARS-CoV-2 hyperimmune serum off-label approved by ANMAT for use according to Regulation 9175/20.
* Pregnant women.
* Lactating women.
* Patients who are on mechanical ventilation or admitted to the ICU at hospital admission.
* Confirmation of another concomitant microbiological cause of pneumonia other than COVID-19

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients younger than 80 years hospitalized at the "Escuela Hogar" Hospital in Corrientes, Argentina, for severe pneumonia diagnosed with SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Mortality at day 28 | 28th day since hospital admission date
  Proportion of patients who die at 28th day since hospital admission date

SECONDARY OUTCOMES:
Mortality at days 14 and 21 after hospital admission. | 14th and 21st days since hospital admission date
  Proportion of patients who die at 14th and 21st days since hospital admission date
Ordinal clinical scale at days 14, 21 and 28 | 14th, 21st and 28th days since hospital admission date
  Proportion of patients in each categorie at 14th, 21st and 28th days since hospital admission
Hospital discharge at days 14, 21 and 28. | 14th, 21st and 28th days since hospital admission date
  Proportion of patients discharged from hospital on days 14, 21 and 28 since hospital admission date
Time to hospital discharge | Time to hospital discharge since hospital admission date in a 28 days follow up period
  Time to hospital discharge since hospital admission date (days).
Patients admitted to Intensive Care Unit. | 28 days follow up period since hospital admission date
  Proportion of patients admitted to Intensive Care Unit in a 28 days follow up period since hospital admission date
Time to discharge from the Intensive Care Unit | 28 days follow up period since hospital admission date
  Time to discharge from the Intensive Care Unit since hospital admission date (days).
Days in Intensive Care Unit. | 28 days follow up period since hospital admission date
  Total days hospitalized in Intensive Care Unit.
Patients on mechanical ventilation | 28 days follow up period since hospital admission date
  Proportion of patients admitted to mechanical ventilation.
Time from the date of hospitalization to the start of mechanical ventilation. | 28 days follow up period since hospital admission date
  Time to mechanical ventilation start since hospital admission date (days).
Adverse events / serious adverse events. | 28 days follow up period since hospital admission date
  Proporcion of participants with adverse events / serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Colonna, Bioch, Principal Investigator — Inmunova S.A.
Locations (1):
- Hospital de Campaña "Escuela Hogar", Corrientes, Argentina